CLINICAL TRIAL: NCT06176664
Title: Oxygen Therapy for Children With Moderate Hypoxemia in Malawi: Pilot Randomized Control Trial
Brief Title: Oxygen Therapy for Children With Moderate Hypoxemia in Malawi
Acronym: NoGoLo2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00421624
Record Dates: First submitted 2023-12-06; First posted 2023-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pneumonia
Keywords: Pneumonia; High flow nasal cannula oxygen; Oxygen; Low and Middle Income Countries; pediatrics
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Pilot trial to assess feasibility of the protocol for a three-armed, open-label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Participants will receive pneumonia care per World Health Organization guidelines. If their oxygen saturation falls below 90% after enrollment, they will be treated with low-flow oxygen.
- Low-flow Oxygen (Experimental): Participants will be treated with low-flow oxygen to achieve a goal oxygen saturation above 94%
  Interventions: Device: Low flow oxygen
- High-flow Nasal Cannula Oxygen (Experimental): Participants will be treated with high-flow nasal cannula oxygen to achieve a goal oxygen saturation above 94%.
  Interventions: Device: High-flow nasal cannula oxygen

INTERVENTIONS:
Device: Low flow oxygen — Standard nasal cannula oxygen up to 2 liters/minute
  Arms: Low-flow Oxygen
Device: High-flow nasal cannula oxygen — High-flow nasal cannula with heating and humidification up to 2 liters/kilogram/minute
  Arms: High-flow Nasal Cannula Oxygen

SUMMARY:
The goal of this pilot clinical trial is to compare standard of care, low-flow oxygen, and high-flow nasal canula oxygen in pediatric patients aged 1-59 months with pneumonia and an oxygen saturation of 90-93% in Malawi. The main question it aims to answer is:

* Does the protocol for the randomized control trial work well?
* Can the researchers safely conduct the protocol for the trial?

Participants will be randomly assigned to one of the three groups (normal care without oxygen, low-flow oxygen, and high-flow nasal cannula oxygen) and treated with that therapy in the hospital. Researchers will look at the ability to safely conduct each part of the study.

DETAILED DESCRIPTION:
Pneumonia is the leading infectious cause of under 5-year-old deaths globally and responsible for >50% of deaths in Africa. The World Health Organization (WHO) defines low blood oxygen saturation (SpO2) levels (hypoxemia) as 90%. Hypoxemia is identified in 31% of child pneumonia cases in Africa and is a key marker of elevated mortality risk. When children are hypoxemic, the WHO recommends oxygen treatment. Importantly, the WHO threshold of 90% for hypoxemia was based on concerns over limited oxygen supply and hospital over-crowding in low- and middle-income countries (LMICs), rather than quality evidence. In most LMICs, low oxygen flow is the mainstay of oxygen delivery. Recently, in high-income settings high-flow nasal cannula (HFNC) oxygen has emerged as a safe and effective alternative. HFNC oxygen delivers higher flow warmed, humidified gas via nasal prongs to reverse hypoxemia, and potentially improve outcomes.

Recent evidence challenges whether the WHO & 90% hypoxemia threshold is optimal for identifying all children at higher risk of mortality in LMICs. One meta-analysis from 13 LMICs reported 3.66-fold-higher odds of death (95% confidence interval (CI), 1.42, 9.47) for children with a SpO2 93%. The investigators research from Malawi and Bangladesh established children with pneumonia and SpO2 between 90-93% (moderate hypoxemia) is common, and, compared to higher SpO2 levels, conveys higher mortality risk. To date, African children with a SpO2 90-93% are not recommended for oxygen treatment. Observational data from Malawi found children with moderate hypoxemia and treated with oxygen had higher survival than those referred with a SpO2 90%. Currently, no randomized trials have determined whether low flow oxygen or HFNC oxygen treatment reduces the mortality of children with moderate hypoxemia (SpO2 90-93%) in African LMICs.

Aim 1: Conduct a pilot open label, three armed, parallel, randomized controlled trial (RCT) comparing standard care, low-flow oxygen, and HFNC oxygen for children with clinical pneumonia and a SpO2 90-93% to determine feasibility of a larger trial. The investigators hypothesize it will be feasible to recruit, randomize, treat, and safely follow-up all participants. Children with SpO2 90-93% will be randomized 1:1:1 to standard care without oxygen (controls), low flow oxygen (intervention #1), or HFNC oxygen (intervention #2). The primary outcome will be feasibility, defined as the proportion of enrolled children with 2 protocol violations. Secondary outcomes include consent refusal, intervention efficacy, participant attrition, and safety.

Aim 2: Determine the prevalence of young Malawian children with a SpO2 90-93% at the designated study hospital. The investigators hypothesize a SpO2 90-93% will be common among children presenting to the trial hospital. The investigators will measure the SpO2 of all children under-five years old (not limited to pneumonia cases) presenting to the hospital 1 week per month over 12-months. Conservatively assuming an average volume of 30 children per day, based on prior data, the investigators will generate 1,400 SpO2 measurements.

ELIGIBILITY:
Inclusion Criteria:

* 1-59 months of age
* Pneumonia (as defined by the World Health Organization)
* Oxygen saturation 90-93% without oxygen

Exclusion Criteria:

* Emergency signs (signs of severe illness as defined by the World Health Organization) including:
* absent or obstructed breathing,
* severe respiratory distress,
* shock,
* decreased mental status,
* convulsions, or
* severe dehydration

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of study protocol as assessed by protocol violations | Enrollment up to 14 days
  Determine overall protocol fidelity, defined as the percentage of enrolled children with < 2 protocol violations, of an open-label, three arm randomized controlled trial comparing low-flow and high-flow nasal cannula (HFNC) oxygen to standard of care without oxygen therapy

SECONDARY OUTCOMES:
Caregiver Trial Acceptability | Day of screening and enrollment
  Determine caregiver trial acceptability, defined as the percentage of caregivers of eligible children who consent to study participation.
Feasibility of screening and enrollment as assessed by percentage of inclusion and exclusion violations | Day of screening and enrollment
  Determine the feasibility of screening and enrollment, defined as the percentage of enrolled children with no inclusion or exclusion criteria violations.
Feasibility of randomization as assessed by percentage of children receiving intervention | 1 hour after randomization
  Determine feasibility of randomization, defined as percentage of children actively receiving the assigned intervention within 1 hours of randomization
Fidelity to treatment failure study definition as assessed by percentage of children with correct treatment failure classification | Enrollment up to 14 days
  Determine fidelity to treatment failure study definition, defined as the percentage of children with a correct treatment failure classification
Fidelity to respiratory supportive care protocol as assessed by percentage of children without a respiratory support protocol violation | Enrollment up to 14 days
  Determine fidelity to respiratory supportive care protocol, defined as the proportion of children without a respiratory support protocol violation
Feasibility of at home follow up as assessed by percentage of participants followed up at home | Enrollment up to 14 days
  Determine feasibility of at home follow up defined as percentage of patients successfully followed up at home with assessment of vital status

OTHER OUTCOMES:
Treatment failure rate | Enrollment up to 14 days
  Determine point estimates and 95% confidence intervals for treatment failure rate for standard of care, conventional low-flow oxygen, and HFNC oxygen arms for children with WHO-defined pneumonia and moderate hypoxemia
Mortality rate | Enrollment up to 14 days
  Determine point estimates and 95% confidence intervals for mortality rate for standard of care, conventional low-flow oxygen, and HFNC oxygen arms for children with WHO-defined pneumonia and moderate hypoxemia
Number of Serious Adverse Events | Enrollment up to 14 days
  Determine point estimate and 95% confidence interval for the rate of serious adverse events (SAEs) for standard of care, conventional low-flow oxygen, and HFNC oxygen arms for children with WHO-defined pneumonia and moderate hypoxemia
Hospital length of stay (days) | Enrollment through hospital discharge up to 30 days
  Determine mean hospital length of stay with standard deviation for standard of care, conventional low-flow oxygen, and HFNC oxygen arms for children with World Health Organization (WHO)-defined pneumonia and moderate hypoxemia

CONTACTS AND LOCATIONS:
Overall Officials: Eric E McCollom, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Salima District Hospital, Salima, Central Region, Malawi

IPD SHARING:
Plan to Share IPD: Yes
The research proposed is a pilot randomized, open-label trial of acute lower respiratory infection with moderate hypoxemia oxygen use in Malawi. The pilot trial will enroll 21 participants with a primary outcome of study feasibility. The datasets will report de-identified patient outcomes including mortality, hospital length of stay, and treatment failure as well as trial feasibility and acceptability data. The shared format of data will be .csv files.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be provided at the time of the primary outcome publication(s) for a period of at least 10 years.
Access Criteria: Publicly shared data will be deposited in an open access repository that meets the specifications required by the NIH. The selected repository will provide metadata, unique identifiers, and data access for at least 10 years. Use of keywords will allow for findability using searches. Access to data will be controlled and limited to qualified investigators who sign a data use agreement and provide a reasonable research question for application to the data. Data requests will require at least a description of the research, objective, design, analysis plan that includes data safeguards, publicly available research use statement, documentation of institutional Review Board (IRB) review and approval. The open access repository will review the request and has final authority for deciding on access to the data. If the study is active, then

REFERENCES:
- [Background] Tortosa F, Izcovich A, Carrasco G, Varone G, Haluska P, Sanguine V. High-flow oxygen nasal cannula for treating acute bronchiolitis in infants: A systematic review and meta-analysis. Medwave. 2021 May 12;21(4):e8190. doi: 10.5867/medwave.2021.04.8190. English, Spanish. PMID 34086669
- [Background] Luo J, Duke T, Chisti MJ, Kepreotes E, Kalinowski V, Li J. Efficacy of High-Flow Nasal Cannula vs Standard Oxygen Therapy or Nasal Continuous Positive Airway Pressure in Children with Respiratory Distress: A Meta-Analysis. J Pediatr. 2019 Dec;215:199-208.e8. doi: 10.1016/j.jpeds.2019.07.059. Epub 2019 Sep 27. PMID 31570155
- [Background] Lin J, Zhang Y, Xiong L, Liu S, Gong C, Dai J. High-flow nasal cannula therapy for children with bronchiolitis: a systematic review and meta-analysis. Arch Dis Child. 2019 Jun;104(6):564-576. doi: 10.1136/archdischild-2018-315846. Epub 2019 Jan 17. PMID 30655267
- [Background] Kawaguchi A, Yasui Y, deCaen A, Garros D. The Clinical Impact of Heated Humidified High-Flow Nasal Cannula on Pediatric Respiratory Distress. Pediatr Crit Care Med. 2017 Feb;18(2):112-119. doi: 10.1097/PCC.0000000000000985. PMID 27741041
- [Background] McKiernan C, Chua LC, Visintainer PF, Allen H. High flow nasal cannulae therapy in infants with bronchiolitis. J Pediatr. 2010 Apr;156(4):634-8. doi: 10.1016/j.jpeds.2009.10.039. Epub 2009 Dec 29. PMID 20036376
- [Background] Moreel L, Proesmans M. High flow nasal cannula as respiratory support in treating infant bronchiolitis: a systematic review. Eur J Pediatr. 2020 May;179(5):711-718. doi: 10.1007/s00431-020-03637-0. Epub 2020 Mar 31. PMID 32232547
- [Background] Hutchings FA, Hilliard TN, Davis PJ. Heated humidified high-flow nasal cannula therapy in children. Arch Dis Child. 2015 Jun;100(6):571-5. doi: 10.1136/archdischild-2014-306590. Epub 2014 Dec 1. PMID 25452315
- [Background] McCollum ED, Mvalo T, Eckerle M, Smith AG, Kondowe D, Makonokaya D, Vaidya D, Billioux V, Chalira A, Lufesi N, Mofolo I, Hosseinipour M. Bubble continuous positive airway pressure for children with high-risk conditions and severe pneumonia in Malawi: an open label, randomised, controlled trial. Lancet Respir Med. 2019 Nov;7(11):964-974. doi: 10.1016/S2213-2600(19)30243-7. Epub 2019 Sep 24. PMID 31562059
- [Background] Chaparro CM, Suchdev PS. Anemia epidemiology, pathophysiology, and etiology in low- and middle-income countries. Ann N Y Acad Sci. 2019 Aug;1450(1):15-31. doi: 10.1111/nyas.14092. Epub 2019 Apr 22. PMID 31008520
- [Background] Allardet-Servent J, Sicard G, Metz V, Chiche L. Benefits and risks of oxygen therapy during acute medical illness: Just a matter of dose! Rev Med Interne. 2019 Oct;40(10):670-676. doi: 10.1016/j.revmed.2019.04.003. Epub 2019 May 1. PMID 31054779
- [Background] McCollum ED, Ahmed S, Roy AD, Chowdhury NH, Schuh HB, Rizvi SJR, Hanif AAM, Khan AM, Mahmud A, Pervaiz F, Harrison M, Reller ME, Simmons N, Quaiyum A, Begum N, Santosham M, Checkley W, Moulton LH, Baqui AH; Projahnmo Study Group in Bangladesh. Effectiveness of the 10-valent pneumococcal conjugate vaccine against radiographic pneumonia among children in rural Bangladesh: A case-control study. Vaccine. 2020 Sep 29;38(42):6508-6516. doi: 10.1016/j.vaccine.2020.08.035. Epub 2020 Aug 29. PMID 32873404
- [Background] Colbourn T, King C, Beard J, Phiri T, Mdala M, Zadutsa B, Makwenda C, Costello A, Lufesi N, Mwansambo C, Nambiar B, Hooli S, French N, Bar Zeev N, Qazi SA, Bin Nisar Y, McCollum ED. Predictive value of pulse oximetry for mortality in infants and children presenting to primary care with clinical pneumonia in rural Malawi: A data linkage study. PLoS Med. 2020 Oct 23;17(10):e1003300. doi: 10.1371/journal.pmed.1003300. eCollection 2020 Oct. PMID 33095763
- [Background] Rahman AE, Hossain AT, Nair H, Chisti MJ, Dockrell D, Arifeen SE, Campbell H. Prevalence of hypoxaemia in children with pneumonia in low-income and middle-income countries: a systematic review and meta-analysis. Lancet Glob Health. 2022 Mar;10(3):e348-e359. doi: 10.1016/S2214-109X(21)00586-6. PMID 35180418
- [Background] McCollum ED, Ginsburg AS. Outpatient Management of Children With World Health Organization Chest Indrawing Pneumonia: Implementation Risks and Proposed Solutions. Clin Infect Dis. 2017 Oct 16;65(9):1560-1564. doi: 10.1093/cid/cix543. PMID 29020216
- [Background] Hooli S, Colbourn T, Lufesi N, Costello A, Nambiar B, Thammasitboon S, Makwenda C, Mwansambo C, McCollum ED, King C. Predicting Hospitalised Paediatric Pneumonia Mortality Risk: An External Validation of RISC and mRISC, and Local Tool Development (RISC-Malawi) from Malawi. PLoS One. 2016 Dec 28;11(12):e0168126. doi: 10.1371/journal.pone.0168126. eCollection 2016. PMID 28030608
- [Background] Hooli S, King C, Zadutsa B, Nambiar B, Makwenda C, Masache G, Lufesi N, Mwansambo C, Malla L, Costello A, Colbourn T, McCollum ED. The Epidemiology of Hypoxemic Pneumonia among Young Infants in Malawi. Am J Trop Med Hyg. 2020 Mar;102(3):676-683. doi: 10.4269/ajtmh.19-0516. PMID 31971153
- [Background] King C, Zadutsa B, Banda L, Phiri E, McCollum ED, Langton J, Desmond N, Qazi SA, Nisar YB, Makwenda C, Hildenwall H. Prospective cohort study of referred Malawian children and their survival by hypoxaemia and hypoglycaemia status. Bull World Health Organ. 2022 May 1;100(5):302-314B. doi: 10.2471/BLT.21.287265. Epub 2022 Mar 25. PMID 35521039
- [Background] Subhi R, Adamson M, Campbell H, Weber M, Smith K, Duke T; Hypoxaemia in Developing Countries Study Group. The prevalence of hypoxaemia among ill children in developing countries: a systematic review. Lancet Infect Dis. 2009 Apr;9(4):219-27. doi: 10.1016/S1473-3099(09)70071-4. PMID 19324294
- [Background] McCollum ED, Bjornstad E, Preidis GA, Hosseinipour MC, Lufesi N. Multicenter study of hypoxemia prevalence and quality of oxygen treatment for hospitalized Malawian children. Trans R Soc Trop Med Hyg. 2013 May;107(5):285-92. doi: 10.1093/trstmh/trt017. PMID 23584373
- [Background] McCollum ED, King C, Hammitt LL, Ginsburg AS, Colbourn T, Baqui AH, O'Brien KL. Reduction of childhood pneumonia mortality in the Sustainable Development era. Lancet Respir Med. 2016 Dec;4(12):932-933. doi: 10.1016/S2213-2600(16)30371-X. Epub 2016 Nov 12. No abstract available. PMID 27843130
- [Background] Lazzerini M, Sonego M, Pellegrin MC. Hypoxaemia as a Mortality Risk Factor in Acute Lower Respiratory Infections in Children in Low and Middle-Income Countries: Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 15;10(9):e0136166. doi: 10.1371/journal.pone.0136166. eCollection 2015. PMID 26372640
- [Background] Walsh BK, Smallwood CD. Pediatric Oxygen Therapy: A Review and Update. Respir Care. 2017 Jun;62(6):645-661. doi: 10.4187/respcare.05245. PMID 28546370
- [Background] Sonego M, Pellegrin MC, Becker G, Lazzerini M. Risk factors for mortality from acute lower respiratory infections (ALRI) in children under five years of age in low and middle-income countries: a systematic review and meta-analysis of observational studies. PLoS One. 2015 Jan 30;10(1):e0116380. doi: 10.1371/journal.pone.0116380. eCollection 2015. PMID 25635911
- [Background] Liu L, Oza S, Hogan D, Chu Y, Perin J, Zhu J, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of under-5 mortality in 2000-15: an updated systematic analysis with implications for the Sustainable Development Goals. Lancet. 2016 Dec 17;388(10063):3027-3035. doi: 10.1016/S0140-6736(16)31593-8. Epub 2016 Nov 11. PMID 27839855